CLINICAL TRIAL: NCT06232174
Title: Study of the Value of Transcutaneous Bilirubin Devices in Jaundiced Newborns at Assiut University Children's Hospital
Brief Title: Value of Transcutaneous Bilirubin Devices
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, marina farah fawzy gad, Pediatric resident, Assiut University
Other Study IDs: transcutaneous bilirubin
Record Dates: First submitted 2024-01-22; First posted 2024-01-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Jaundice
Keywords: Neonatal jaundice
MeSH Terms: conditions — Jaundice; Jaundice, Neonatal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 25 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to compare the value of transcutaneous bilirubin devices versus serum bilirubin in jaundiced neonates

DETAILED DESCRIPTION:
Neonatal jaundice, commonly found in 60% of normal newborns, is normally a self-resolving episode ending 72 to 96 h after birth. Transient elevation of blood bilirubin occurs by combination of an increase in red blood cell destruction and concomitant decrease in hepatic bilirubin conjugation. (1) Visible jaundice is present in most term and near-term newborns during the first week of life. Although it is mostly a benign condition, healthcare professionals should keep in mind rare but severe adverse outcomes of serious hyperbilirubinemia (2). Newborn infants must be monitored to identify those who might develop severe hyperbilirubinemia and, in rare cases, acute bilirubin encephalopathy or kernicterus.Kernicterus is associated with a high mortality rate and survivors usually suffer from complications such as athetoid cerebral palsy, highfrequency hearing loss and intellectual disability(3).

Severe neonatal hyperbilirubinemia and its sequelae can be prevented with appropriate serum bilirubin monitoring and early treatment involving phototherapy or exchange blood transfusion (4). In the 2004 American Academy of Pediatrics Subcommittee on Hyperbilirubinemia guideline, total serum bilirubin (TSB) or transcutaneous bilirubin (TcB) measurement is recommended before discharge from the maternity hospital to evaluate the risk of subsequent severe hyperbilirubinemia in all newborns (5). To measure bilirubin levels, the total serum bilirubin (TSB) measured by the biochemical laboratory is still considered a gold standard, but it is invasive, requiring needle pricks that carry the risk for iatrogenic anemia, puncture site infection, bacteremia, and osteomyelitis, and cause pain and stress to the neonates(6). The turn around time for bilirubin test results may delay the initiation of therapy for neonatal hyperbilirubinemia. In recent years, the transcutaneous bilirubinometer, which uses photometry to detect bilirubin levels, has been used as an alternative to estimate the bilirubin levels(4). TcB meters estimate total serum or plasma bilirubin using multiwave length spectral reflection from the skin surface.(7) Transcutaneous bilirubinometry (TcB) developed due to several converging influences and factors as the recognition that yellow skin color is due to the deposition of bilirubin,1 a chromophore molecule that, with advancements in optical science, could be quantitatively measured(8). Transcutaneous bilirubinometry (TcB) has the following advantages ease of use, non-invasive nature and reduction in the number of inpatient TSB determinations reduced expense when compared to a serum bilirubin, immediate results, and superior performance over visual assessment of jaundice. The first attempt at non-invasive measurement of bilirubin goes back to the 1960's when the icterometer was introduced. This device, based on reflectance, had poor analytical specificity and sensitivity, and poor reproducibility with coefficient of variations ranging between 20 and 40%. In the past years, bilirubinometers have gradually been improved and are now based on simultaneous multiple wavelength analysis (9)

ELIGIBILITY:
Inclusion Criteria:

* They were born between 35 and 42 weeks of gestation, had a birth weight of more than 2 kg, and were aged between 0 days and 28 days

Exclusion Criteria:

* Exclusion criteria are severely ill neonates, neonates with a lethal congenital malformation, and or had skin disease, had received phototherapy before, and received exchange transfusion.

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: jaundiced neonates followed in assiut university children's hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
diagnostic accuracy of transcutaneous bilirubin devices as a diagnostic test for hyperbilirubinaemia in newborns | 20 days
  diagnostic test accuracy studies comparing TcB and TsB measurement for hyperbilirubinaemia in newborns

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Gamil, Professor, Study Director — Assiut University
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Carceller-Blanchard A, Cousineau J, Delvin EE. Point of care testing: transcutaneous bilirubinometry in neonates. Clin Biochem. 2009 Feb;42(3):143-9. doi: 10.1016/j.clinbiochem.2008.09.106. Epub 2008 Oct 2. PMID 18929553
- [Background] Bhutani VK, Stark AR, Lazzeroni LC, Poland R, Gourley GR, Kazmierczak S, Meloy L, Burgos AE, Hall JY, Stevenson DK; Initial Clinical Testing Evaluation and Risk Assessment for Universal Screening for Hyperbilirubinemia Study Group. Predischarge screening for severe neonatal hyperbilirubinemia identifies infants who need phototherapy. J Pediatr. 2013 Mar;162(3):477-482.e1. doi: 10.1016/j.jpeds.2012.08.022. Epub 2012 Oct 5. PMID 23043681
- [Background] Ministry of Health Malaysia. Clinical practice guidelines: management of neonatal jaundice. 2nd ed. Kuala Lumpur, Malaysia: Ministry of Health; 2014.
- [Background] Mohamed M, Ibrahim NR, Ramli N, Abdul Majid N, Yacob NM, Nasir A. Comparison between the Transcutaneous and Total Serum Bilirubin Measurement in Malay Neonates with Neonatal Jaundice. Malays J Med Sci. 2022 Feb;29(1):43-54. doi: 10.21315/mjms2022.29.1.5. Epub 2022 Feb 23. PMID 35283687
- [Background] American Academy of Pediatrics Subcommittee on Hyperbilirubinemia. Management of hyperbilirubinemia in the newborn infant 35 or more weeks of gestation. Pediatrics. 2004 Jul;114(1):297-316. doi: 10.1542/peds.114.1.297. PMID 15231951
- [Background] Taylor JA, Burgos AE, Flaherman V, Chung EK, Simpson EA, Goyal NK, Von Kohorn I, Dhepyasuwan N; Better Outcomes through Research for Newborns Network. Discrepancies between transcutaneous and serum bilirubin measurements. Pediatrics. 2015 Feb;135(2):224-31. doi: 10.1542/peds.2014-1919. Epub 2015 Jan 19. PMID 25601981
- [Background] Hussain AS, Shah MH, Lakhdir M, Ariff S, Demas S, Qaiser F, Ali SR. Effectiveness of transcutaneous bilirubin measurement in managing neonatal jaundice in postnatal ward of a tertiary care hospital in Pakistan. BMJ Paediatr Open. 2017 Aug 31;1(1):e000065. doi: 10.1136/bmjpo-2017-000065. eCollection 2017. PMID 29637112
- [Background] Engle WD, Jackson GL, Engle NG. Transcutaneous bilirubinometry. Semin Perinatol. 2014 Nov;38(7):438-51. doi: 10.1053/j.semperi.2014.08.007. Epub 2014 Oct 3. PMID 25282473
- [Background] GOSSET IH. A perspex icterometer for neonates. Lancet. 1960 Jan 9;1(7115):87-8. doi: 10.1016/s0140-6736(60)92902-0. No abstract available. PMID 13851385